CLINICAL TRIAL: NCT00668083
Title: Observational Retrospective Trial on Sequential Hormonal Therapy in Patients
Brief Title: Observational Retrospective Trial on Sequential Hormonal Therapy in Patients With Prostate Cancer
Acronym: Sorse
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Italy: Ethics Committee, AstraZeneca
Other Study IDs: NIS-OIT-CAS-2007/1
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Prostate Cancer
Keywords: second line; Prostate Cancer; bicalutamide; biochemical relapse/progression in patients with Prostate Cancer treated with bicalutamide 150mg
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational Retrospective trial on sequential hormonal therapy in patients with Prostate Cancer

ELIGIBILITY:
Inclusion Criteria:

* non metastatic Prostate Cancer
* previous treatment with bicalutamide 150mg
* biochemical relapse/progression

Exclusion Criteria:

* use of other treatments for Prostate Cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: THIS IS A RETROSPECTIVE TRIAL THEREFORE CLINICAL DATA ARE FROM ARCHIVED CLINICAL RECORD OF PATIENTS WHO WERE ADMITTED IN THE HOSPITAL.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Estimated)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Hormonal sensitivity to second line treatment for CaP after Bicalutamide | six months

SECONDARY OUTCOMES:
median duration of second and third line treatments; | six months

CONTACTS AND LOCATIONS:
Overall Officials: Davide Meani, MD, Study Director — AstraZeneca Medical Dept
Locations (12):
- Italy (12):
  - Research Site, Acquaviva delle Fonti
  - Research Site, Ancona
  - Research SIte, Florence
  - Research Site, Matera
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Portogruaro
  - Research Site, Roma
  - Research Site, Viareggio